CLINICAL TRIAL: NCT07355010
Title: A Randomized, Open-label, Double-cohort Study of Fluzoparib Combined With Famitinib Malate or SHR-1701 for Neoadjuvant Therapy in Patients With Advanced Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qinglei Gao (Other)
Responsible Party: Sponsor-Investigator, Qinglei Gao, doctor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-OC-II-016
Record Dates: First submitted 2025-11-16; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — famitinib; SHR-1701

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fuzuloparib and Famitinib (Experimental): fuzuloparib and famitinib
  Interventions: Drug: fuzuloparib; Drug: Famitinib
- Fuzuloparib and SHR-1701 (Experimental): fuzuloparib and SHR-1701
  Interventions: Drug: fuzuloparib; Drug: SHR-1701

INTERVENTIONS:
Drug: fuzuloparib — fuzuloparib 150mg bid PO
Drug: Famitinib — famitinib 10mg qd PO
  Arms: Fuzuloparib and Famitinib
Drug: SHR-1701 — SHR-1701 1800 mg IV Q3W
  Arms: Fuzuloparib and SHR-1701

SUMMARY:
This study is a randomized, open-label, double-cohort, national multi-center clinical research. The aim is to evaluate the newly diagnosed FIGO 2014 stage III-IV pathology of neoadjuvant therapy with fluzoparib combined with famitinib or fluzoparib combined with SHR-1701, based on the Fagotti laparoscopy score or upper abdominal Suidan's by the researchers The CT score assesses the efficacy and safety of patients with germline BRCA wild-type ovarian cancer who cannot achieve R0 resection or cannot tolerate initial cytoreductive surgery, as well as the efficacy and safety of surgery, adjuvant therapy, and combined maintenance treatment regimens based on fluzoparib.

The primary endpoint was the objective response rate (ORR) after neoadjuvant therapy as assessed by the researchers based on the RECIST v1.1 criteria. Meanwhile, the chemotherapy response score (CRS), event-free survival (EFS), disease-free survival (DFS), progression-free survival (PFS), and overall survival (OS) were also examined. The safety, tolerability and patient-reported outcomes (EQ-5D-5L) of the two cohorts were investigated.

A total of 104 newly diagnosed epithelial ovarian cancer patients with germline BRCA wild-type (FIGO 2014 stage III-IV) are planned to be enrolled.

ELIGIBILITY:
Inclusion criteria：

* The subjects voluntarily joined this study and signed the informed consent form;
* Age ≥18 years old (calculated from the date of signing the informed consent);
* Newly diagnosed high-grade (or moderately and poorly differentiated) serous ovarian cancer, fallopian tube cancer or primary peritoneal cancer in pathology; Ovarian endometrioid adenocarcinoma of grade ≥ II; Mixed tumor: High-grade serous type or ≥ grade II endometrioid components must be present.
* FIGO 2014 Phase III-IV;
* The subjects have at least one measurable lesion that can be evaluated by CT or MRI (RECIST v1.1) ;
* After assessment by the researcher, R0 resection cannot be achieved or the surgery cannot be tolerated;

The criteria for judging that <s:1> cannot reach R0 resection include:

1. Fagotti endoscopic score ≥8 points;
2. When laparoscopic assessment methods are difficult to implement, an upper abdominal Suidan's CT score of ≥3 points can be adopted.

The criteria for the inability to tolerate surgery may be considered:

1. Body Mass Index: BMI≥40;
2. Multiple chronic diseases;
3. Malnutrition or hypoproteinemia;
4. Moderate to massive ascites;
5. Newly diagnosed venous thromboembolism;
6. Physical condition: ECOG PS > 2;
7. Other reasons as determined by the researcher;

   * ECOG PS: 0-2;
   * The subject has been tested and confirmed by a professional institution to be of the wild type of germline BRCA1/2.
   * The functions of vital organs meet the following requirements (no blood components or cell growth factors are allowed to be used within 14 days before the first administration) :

<s:1> Absolute neutrophil count ≥1.5×109/L; <s:1> platelet count ≥100×109/L; <s:1> hemoglobin ≥9 g/dL; Serum albumin ≥3g/dL; Bilirubin ≤1.5 times ULN; <s:1> ALT and AST ≤2.5 times ULN, and ≤5 times ULN in the presence of liver metastasis; Serum creatinine ≤1.5 times ULN, or creatinine clearance ≥60 mL/min (calculated according to the Cockcroft-Gault formula);

* Fertile subjects must undergo a blood pregnancy test with a negative result within one week before the first administration of the drug, and must not be in the lactation period. They must agree to take effective contraceptive measures during the trial period and for six months after the last administration of the trial drug. If there is any suspected or confirmed pregnancy, they must immediately notify the investigator.
* The subjects were willing to cooperate in completing the questionnaire survey on quality of life during the trial treatment and follow-up, and agreed that the results of the questionnaire survey could be used for clinical research.

Exclusion criteria：

* In the past (within 5 years) or concurrently with other uncured malignant tumors, for cured thyroid cancer, basal cell carcinoma of the skin, carcinoma in situ, and those who have completed radical mastectomy > Breast cancer that has not recurred for three years is excluded.
* The subjects have untreated central nervous system metastases Patients who have previously received systemic or radical treatment for brain or meningeal metastases (radiotherapy or surgery), and whose stability has been maintained for at least one month as confirmed by imaging, and who have stopped systemic hormone therapy (10mg/ day prednisone or other equivalent therapeutic hormones) for more than two weeks and have no clinical symptoms, can be included.
* The subjects have previously received treatment with known or possible PARP inhibitors, anti-angiogenic drugs, and PD-L1/TGF-β.
* Those who are unable to swallow tablets normally or have abnormal gastrointestinal function, which the researcher determines may affect drug absorption;
* Those who have experienced intestinal obstruction or gastrointestinal perforation in the recent period (within 3 months);
* There are poorly controlled clinical symptoms or diseases of the heart, such as: (1) NYHA grade 2 or above heart failure; (2) unstable angina pectoris; (3) Myocardial infarction occurred within one year; (4) clinically significant supventricular or ventricular arrhythmias requiring treatment or intervention; (5) QTc> 470ms;
* If any severe bleeding event with a grade of 2 or above in CTCAE 5.0 occurs within 4 weeks before the first medication, such as gastrointestinal bleeding, hemorrhagic gastric ulcer or phlebitis, etc., and the fecal occult blood is positive during the baseline period, a re-examination can be conducted. If the re-examination is still positive, a gastroscopy or colonoscopy should be performed in combination with clinical judgment when necessary.
* The subject has received platelet or red blood cell transfusion within 14 days before the start of treatment;
* Accompanied by active ulcers, unhealed wounds or fractures;
* The subjects had active infections or developed unexplained fever during the screening period or before the first administration. 38.5 degrees
* The subject has congenital or acquired immune deficiency (such as HIV infection), or active hepatitis (Hepatitis B reference: HBsAg positive and HBV DNA≥500 IU/ml or 1000 copies/mL; Hepatitis C reference: HCV antibody positive and HCV RNA > upper limit of normal value);
* Those who had previously received radiotherapy, chemotherapy, hormone therapy, or molecular targeted therapy and had less than 4 weeks before the completion of the treatment (the last medication) (for oral molecular targeted drugs, it was less than 5 drug half-lives); Adverse events caused by previous treatment (excluding alopecia) have not recovered to grade ≤1 (CTCAE 5.0);
* Within 6 months prior to the first medication, there have been events of grade ≥3 arterial thrombosis or venous thrombosis, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.
* Those with a history of hereditary or acquired bleeding or coagulation disorders (such as hemophilia patients, coagulation disorders, thrombocytopenia, etc.);
* During the study period, the subjects may receive other systemic anti-tumor treatments;
* Those with hypertension who have not achieved good control through antihypertensive drug treatment (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
* The subjects are pregnant, breastfeeding or plan to become pregnant during the study treatment period;
* As determined by the researchers, the subjects have other factors that may lead to the forced termination of this study, such as other serious diseases (including mental illness) requiring combined treatment, severe laboratory test abnormalities, accompanied by family or social factors that may affect the safety of the subjects, or the collection of data and samples.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate，ORR | From enrollment to the end of neoadjuvant treatment at around 8 weeks"

SECONDARY OUTCOMES:
event free survival | It is defined as the time from the start of randomization to the first occurrence of any of the following events (disease progression beyond surgical treatment, local or distant recurrence, death of any cause), whichever occurs first, up to 5 years.
disease free survival | It is defined as the period from the first study medication in the adjuvant therapy stage after cytoreductive surgery to disease recurrence or death due to any cause (whichever occurs first), up to 5 years.
progression free survival | It is defined as the period from the start of the first study medication in the maintenance treatment stage to tumor progression or death for any reason (whichever occurs first), up to 5 years.

IPD SHARING:
Plan to Share IPD: No